CLINICAL TRIAL: NCT04167930
Title: The Analysis for Factors Affecting Termination of Treatment and Treatment Satisfaction of Korean Medicine in Traffic Accident Injury Patients: A Retrospective Study With Survey
Brief Title: The Analysis for Termination of Treatment and Satisfaction in Traffic Accident Patient
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Other Study IDs: JS-CT-2019-07
Record Dates: First submitted 2019-11-11; First posted 2019-11-19 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Accidents, Traffic; Whiplash Injuries
Keywords: traffic accident; traditional Korean medicine; car insurance; whiplash injury
MeSH Terms: conditions — Whiplash Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: electronic medical record(EMR) Data and patient survey — 1. Retrospective Data Collection (1) Neck Disability Index (NDI), Oswestry Low Back Disability Index(ODI), euroqol-5 dimension(EQ-5D) scores during hospitalization (2) symptom onset date, symptom onset motive, past history, accident occurrence date, accident treatmen termination agreement date, etc.
  2. Question items (consistent with the case record) according to the purpose of the investigation (1) General: Demographic sociological characteristics (gender, age, occupation, income, etc.) (2) Matters concerning the correlation between traffic accident agreements and symptoms

SUMMARY:
Data of one hospital will be used to find out the patient's satisfaction with the treatment, analyze the factors effecting on the treatment termination.

Also, plan to see if there is a correlation between prognosis according to the seriousness of the accident. In addition, investigators want to find out the participants' perception of car insurance and their satisfaction with traditional Korean medicine treatment.

DETAILED DESCRIPTION:
Retrospective data will be extracted using electronic medical records and computerized data of hospitalized patients. Based on this, investigators will conduct research in the form of prospective survey and analyze the causal relationship and factors using the two data.

The hospital's medical records will be used to analyze the patient's condition during the hospitalization period and to determine the situation after the end of treatment through questionnaire. The questionnaire will be developed after consultation with experts from musculoskeletal system and related societies, and will be used for the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 65
* A traffic accident injury patient who had been hospitalized at Haeundae Jaseng Korean Medicine Hospital from Jan. 01, 2016 to Dec. 31, 2018.

Exclusion Criteria:

* People whose traffic accidents are not yet agreed to
* Those who have not exceeded 90 days (3 months) since the conclusion of the agreement
* Persons unable to communicate

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who ended up the hospitalization and treatment through car insurance in Haeundae Jaseng Korean Medicine Hospital
Sampling Method: Non-Probability Sample
Enrollment: 682 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Pain duration after treatment termination | Finish all survey by Nov 2019
  duration will be checked in week
Spent treatment fee after agreement with car insurance | Finish all data collection by Nov 2019
  fee will be measured in tens of thousands

SECONDARY OUTCOMES:
Change in Neck Disability Index (NDI) | Finish all data collection by Nov 2019
  Neck Disability Index (NDI) scores during hospitalization
Change in Oswestry Disability Index (ODI) | Finish all data collection by Nov 2019
  Oswestry Disability Index (ODI) scores during hospitalization
Change in EuroQol 5-dimensions 5-levels | Finish all data collection by Nov 2019
  EuroQol 5-dimensions 5-levels scores during hospitalization
situation of of traffic accident | Finish all survey by Nov 2019
  Whether in car traffic accident or out car traffic accident
Numeric rating scale (NRS) score | Finish all survey by Nov 2019
  pain score at the accident time
Whiplash-associated disorder (WAD) grade. | Finish all survey by Nov 2019
  seriousness of accidents
overall condition of patient after treatment termination | Finish all survey by Nov 2019
  After the termination of the treatment, confirm that additional treatment was carried out using private expenses and reconfirm the pain after the termination of the treatment.
satisfaction of car insurance | Finish all survey by Nov 2019
  Patients' satisfaction questionnaire (0~10 score) 10 is better
Satisfaction with Korean medicine treatment for traffic accident injury | Finish all survey by Nov 2019
  Patients' satisfaction questionnaire (0~10 score), 10 is better

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Study Chair — Jaseng Medical Foundation
Locations (1):
- Haeundae Jaseng Hospital of Korean Medicine, Busan, South Korea